CLINICAL TRIAL: NCT06160765
Title: The Efficacy of High Density Formula1.5 kcal/ml or 1 kcal/ml On Catch Up Growth In Growth Faltering Children With Feeding Difficulties
Brief Title: The Efficacy of High Density Formula 1.5 kcal/ml or 1 kcal/ml On Catch Up Growth In Growth Faltering Children
Status: Completed | Type: Observational
Sponsor: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Nur Aisiyah Widjaja, Principal Investigator on Nutrition and Metabolic Disease, Universitas Airlangga
Other Study IDs: High Density Formula; UA number (Other: Airlangga University)
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Growth Faltering; High Density Formula; Catch Up Growth
Keywords: Growth Failure; Growth Faltering; High Density Formula; Catch Up Growth
MeSH Terms: conditions — Failure to Thrive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1.5 kcal/ml High Density Formula: This group consist of patients who are able to consume 300-400 kcal of solid food and given 400 cc High Density Formula 1.5 kcal/ml equivalent to 600 kcal
- 1 kcal/ml High Density Formula: This group consist of patients who are able to consume 500-600 kkal of solid food and given 400 cc High Density Formula 1 kcal/ml equivalent to 400 kcal

SUMMARY:
High density calorie is an Oral Nutrition Supplement (ONS) which is a high calorie formula (High Density Formula) and suggested as nutritional therapy to assist children who are undernourished or undergoing growth faltering. The World Health Organization (WHO) and the Indonesian Ministry of Health have established regulations governing the use of ONS for children suffering from undernutrition, whether or not an infection is present. ONS available on the Indonesian market provides an energy density of between 1-1.5 kcal/ml.

This study has the potential to clarify the advantages of ONS administration and evaluate its efficacy in comparison to nutritional therapy (1 kcal/ml or 1.5 kcal/ml) to facilitate rapid catch-up growth by examining the rate of increase in body weight, body lenght and undernourished children, particularly when infection is present.

Purposes:

1. Analyze the effect of the 1.5 kcal/ml high dense formula (ONS) on the average weight gain in undernourished children accompanied by infections
2. Analyze the effect of the 1.5 kcal/ml calorie dense formula (ONS) on the average increase in PB in undernourished children accompanied by infections
3. Analyze the effect of the 1 kcal/ml calorie dense formula (ONS) on the average weight gain in undernourished children accompanied by infections
4. Analyze the effect of 1 kcal/ml calorie dense formula (ONS) on the average increase in PB in undernourished children accompanied by infections
5. Analyze the effect of the 1.5 kcal/ml calorie dense formula (ONS) on changes in nutritional status in undernourished children accompanied by infections

DETAILED DESCRIPTION:
This research is a retrospective observational study using medical record data from the EMR Husada Utama Hospital. Based on the EMR, data will be taken on patients who are able to consume 300-400 kcal of solid food, given 400 cc ONS 1.5 kkal/ml (Nutrini drink) equivalent to 600 kcal as group 1. Patients who are able to consume 500-600 kcal solid food are given 1 kkal/ml 400 cc ONS (SGM optigrow) equivalent 400 kcal as group 2. The rate of increase body weight and body height will be measured at day 0, 30 , 60 and 90 after consumed high dense formula, then it will be plotted in WHO Growth Chart to show the enhancement of nutrition status.

The statistical analysis including test of normality and homogeneity test, followed by paired sample T-test or Wilcoxon, depend on the normality and homogeneity test.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 years - 5 years, are diagnosed tuberculosis (TB) and urinary tract infection (UTI)
* Children who have feeding difficulties
* Children who malnourished or have undergoing weight malnutrition

Exclusion Criteria:

* Children with fluid retention
* Children with organomegaly
* Children with tumor masses.
* Children with congenital abnormalities
* Children wither cerebral palsy, hormonal disorders, and syndromes.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study collect EMRs of private patients at the outpatient pediatric clinic at the Husada Utama Hospital, with a range of November 2021-November 2023 who met the inclusion and exclusion criteria to reach the desired population
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Body Weight | 3 months
  Body weight will be measured using Tanita RD 953-BK digital scale (presenting in mean +/- SD, in kg). The subjects were asked to step at the scale in an upright state. The body weight appears on the screen and is then noted in the data collection sheet. The subject must use light clothes without accessories or footwear
Body Height | 3 months
  Body height will be measured using Seca 213 stadiometer. The subjects were asked to step at the stadiometer base in an upright state, with the heel, the buttock, and the shoulder blade touching the scale pool. The chin up, look straight ahead. The head slider was lowered until it touches the cranium. Noted the body height in the data collection sheet (presenting in mean +/- SD, in cm). The subject must use light clothes without accessories or footwear, such as hats or hair ponytail.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Aisiyah Widjaja, Ph.D, Principal Investigator — Child Health Department, Faculty of Medicine, Universitas Airlangga
Locations (1):
- Husada Utama Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maleta K. Undernutrition. Malawi Med J. 2006 Dec;18(4):189-205. No abstract available. PMID 27529011
- [Background] Zhang Z, Li F, Hannon BA, Hustead DS, Aw MM, Liu Z, Chuah KA, Low YL, Huynh DTT. Effect of Oral Nutritional Supplementation on Growth in Children with Undernutrition: A Systematic Review and Meta-Analysis. Nutrients. 2021 Aug 30;13(9):3036. doi: 10.3390/nu13093036. PMID 34578914
- [Background] Thomson KH, Rice S, Arisa O, Johnson E, Tanner L, Marshall C, Sotire T, Richmond C, O'Keefe H, Mohammed W, Raffle A, Hanratty B, McEvoy CT, Craig D, Ramsay SE. Effectiveness and cost-effectiveness of oral nutritional supplements in frail older people who are malnourished or at risk of malnutrition: a systematic review and meta-analysis. Lancet Healthy Longev. 2022 Oct;3(10):e654-e666. doi: 10.1016/S2666-7568(22)00171-4. Epub 2022 Sep 15. PMID 36116457
- [Background] Pedrianes-Martin PB, Dassen-de-Monzo C, Guardia-Baena JM, Riestra-Fernandez M, Salom-Vendrell C, PerceptiONS Group, Calvo-Barbero A, Lizan-Tudela L. Physicians' Perception of Oral Nutritional Supplement Acceptance and Tolerability in Malnourished Outpatients: PerceptiONS Study. Nutrients. 2023 Feb 28;15(5):1219. doi: 10.3390/nu15051219. PMID 36904218
- [Background] Devaera Y, Syaharutsa DM, Jatmiko HK, Sjarif DR. Comparing Compliance and Efficacy of Isocaloric Oral Nutritional Supplementation Using 1.5 kcal/mL or 1 kcal/mL Sip Feeds in Mildly to Moderately Malnourished Indonesian Children: A Randomized Controlled Trial. Pediatr Gastroenterol Hepatol Nutr. 2018 Oct;21(4):315-320. doi: 10.5223/pghn.2018.21.4.315. Epub 2018 Oct 10. PMID 30345245
- [Background] Stratton RJ, Elia M. Encouraging appropriate, evidence-based use of oral nutritional supplements. Proc Nutr Soc. 2010 Nov;69(4):477-87. doi: 10.1017/S0029665110001977. Epub 2010 Aug 10. PMID 20696091
- [Background] Ui Dhuibhir P, Collura N, Walsh D. Complete Oral Nutritional Supplements: Dietitian Preferences and Clinical Practice. J Diet Suppl. 2019;16(1):40-50. doi: 10.1080/19390211.2018.1428260. Epub 2018 Mar 9. PMID 29521557
- [Background] Hubbard GP, Fry C, Sorensen K, Casewell C, Collins L, Cunjamalay A, Simpson M, Wall A, Van Wyk E, Ward M, Hallowes S, Duggan H, Robison J, Gane H, Pope L, Clark J, Stratton RJ. Energy-dense, low-volume paediatric oral nutritional supplements improve total nutrient intake and increase growth in paediatric patients requiring nutritional support: results of a randomised controlled pilot trial. Eur J Pediatr. 2020 Sep;179(9):1421-1430. doi: 10.1007/s00431-020-03620-9. Epub 2020 Mar 13. PMID 32170451
- [Background] Loman BR, Luo M, Baggs GE, Mitchell DC, Nelson JL, Ziegler TR, Deutz NE, Matarese LE; NOURISH Study Group. Specialized High-Protein Oral Nutrition Supplement Improves Home Nutrient Intake of Malnourished Older Adults Without Decreasing Usual Food Intake. JPEN J Parenter Enteral Nutr. 2019 Aug;43(6):794-802. doi: 10.1002/jpen.1467. Epub 2018 Nov 22. PMID 30565718
- [Background] Adu-Afarwuah S, Lartey A, Brown KH, Zlotkin S, Briend A, Dewey KG. Randomized comparison of 3 types of micronutrient supplements for home fortification of complementary foods in Ghana: effects on growth and motor development. Am J Clin Nutr. 2007 Aug;86(2):412-20. doi: 10.1093/ajcn/86.2.412. PMID 17684213